CLINICAL TRIAL: NCT01153269
Title: Long-term Effectiveness and Safety in Hepatitis-co-infected Patients
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: KAL 1 HO
Record Dates: First submitted 2010-02-26; First posted 2010-06-30 (Estimated); Results first posted 2011-12-19 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-11

CONDITIONS: Human Immunodeficiency Virus-Infection
Keywords: Human Immunodeficiency Virus; Co-infection with Hepatitis B or Hepatitis C; Tolerability; Effectiveness
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hepatitis C | interventions — Lopinavir; Ritonavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV-infected patients with hepatitis co-infection: HIV-infected patients with co-infections of Hepatitis B or Hepatitis C
  Interventions: Drug: Lopinavir/Ritonavir (Kaletra)

INTERVENTIONS:
Drug: Lopinavir/Ritonavir (Kaletra) — 3 capsules 2xdaily or 2 tablets 2xdaily Kaletra

SUMMARY:
The aim of the study is to observe the tolerability and effectiveness of Kaletra in Human Immunodeficiency Virus/Hepatitis-B Virus and Human Immunodeficiency Virus/Hepatitis-C Virus co-infected patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients infected by HIV-1 and HBV or HCV
* Age ≥18 years
* Patients who were initiated on a LPV/r containing antiretroviral (ARV) regimen

Exclusion Criteria:

- Contraindications as described in SmPC (summary of product characteristics) at the time of prescription

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample, Human Immunodeficiency Virus-infected patients with Hepatitis B or C co-infections
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2001-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Simianer, MD, Study Director — Abbott Germany, Medical Department
Locations (8):
- Germany (8):
  - Site Reference ID/Investigator# 27575, Berlin
  - Site Reference ID/Investigator# 27592, Berlin
  - Site Reference ID/Investigator# 27588, Dortmund
  - Site Reference ID/Investigator# 27583, Frankfurt
  - Site Reference ID/Investigator# 27587, Frankfurt
  - Site Reference ID/Investigator# 27607, Hamburg
  - Site Reference ID/Investigator# 5355, Krefeld
  - Site Reference ID/Investigator# 27604, Münster

RESULTS

PARTICIPANT FLOW:
Groups:
- HIV-infected Participants With Hepatitis Co-infection: HIV-infected participants with co-infections of hepatitis B or hepatitis C.
Period: Overall Study
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Started | 33
Participants Analyzed | 33
Completed | 31
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Antiretroviral therapy break | 1

BASELINE CHARACTERISTICS:
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Number analyzed (Participants) | 33
Age Continuous [Mean (Standard Deviation); unit: years] | 42.4 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 25
Region of Enrollment [Number; unit: participants]
  Germany | 33
Hepatitis Co-infection [Number; unit: participants] — The number of participants with hepatitis B or hepatitis C co-infection.
  participants
    Chronic hepatitis B | 9
    Chronic hepatitis C | 24
Duration of HIV infection [Mean (Standard Deviation); unit: years] — How long participants had been diagnosed with HIV infection at Baseline. Based on 32 participants.
  years | 9.7 (7.4)

OUTCOME MEASURES:

1. Primary Outcome: Aspartate Aminotransferase (AST) / Alanine Aminotransferase (ALT) Parameters
Description: The decision to perform aspartate aminotransferase (AST) and alanine aminotransferase (ALT) laboratory tests to monitor participants' liver function was left to the treating physician's clinical judgment. The mean values and standard deviations for those tested at Baseline are presented.
Time Frame: Baseline
Population: Participants with aspartate aminotransferase and alanine aminotransferase results at Baseline.
Measure: Mean (Standard Deviation); unit: U/liter
Groups:
- HIV-infected Participants With Hepatitis Co-infection: AST: Aspartate aminotransferase (AST) results for HIV-infected participants with hepatitis B or hepatitis C co-infection.
- HIV-infected Participants With Hepatitis Co-infection: ALT: Alanine aminotransferase (ALT) results for HIV-infected participants with hepatitis B or hepatitis C co-infection.
Arm/Group | HIV-infected Participants With Hepatitis Co-infection: AST | HIV-infected Participants With Hepatitis Co-infection: ALT
Number analyzed (Participants) | 25 | 24
U/liter | 64 (63) | 69 (88)

2. Primary Outcome: Aspartate Aminotransferase (AST) / Alanine Aminotransferase (ALT) Parameters
Description: The decision to perform aspartate aminotransferase (AST) and alanine aminotransferase (ALT) laboratory tests to monitor participants' liver function was left to the treating physician's clinical judgment. The mean values and standard deviations for those tested at Week 4 are presented.
Time Frame: Week 4
Population: Participants with aspartate aminotransferase and alanine aminotransferase results at Week 4.
Measure: Mean (Standard Deviation); unit: U/liter
Arm/Group | HIV-infected Participants With Hepatitis Co-infection: AST | HIV-infected Participants With Hepatitis Co-infection: ALT
Number analyzed (Participants) | 26 | 26
U/liter | 85 (96) | 85 (86)

3. Primary Outcome: Aspartate Aminotransferase (AST) / Alanine Aminotransferase (ALT) Parameters
Description: The decision to perform aspartate aminotransferase (AST) and alanine aminotransferase (ALT) laboratory tests to monitor participants' liver function was left to the treating physician's clinical judgment. The mean values and standard deviations for those tested at Week 12 are presented.
Time Frame: Week 12
Population: Participants with aspartate aminotransferase and alanine aminotransferase results at Week 12.
Measure: Mean (Standard Deviation); unit: U/liter
Arm/Group | HIV-infected Participants With Hepatitis Co-infection: AST | HIV-infected Participants With Hepatitis Co-infection: ALT
Number analyzed (Participants) | 23 | 24
U/liter | 69 (50) | 85 (79)

4. Primary Outcome: Aspartate Aminotransferase (AST) / Alanine Aminotransferase (ALT) Parameters
Description: The decision to perform aspartate aminotransferase (AST) and alanine aminotransferase (ALT) laboratory tests to monitor participants' liver function was left to the treating physician's clinical judgment. The mean values and standard deviations for those tested at Week 24 are presented.
Time Frame: Week 24
Population: Participants with aspartate aminotransferase and alanine aminotransferase results at Week 24.
Measure: Mean (Standard Deviation); unit: U/liter
Arm/Group | HIV-infected Participants With Hepatitis Co-infection: AST | HIV-infected Participants With Hepatitis Co-infection: ALT
Number analyzed (Participants) | 23 | 23
U/liter | 78 (94) | 97 (134)

5. Primary Outcome: Aspartate Aminotransferase (AST) / Alanine Aminotransferase (ALT) Parameters
Description: The decision to perform aspartate aminotransferase (AST) and alanine aminotransferase (ALT) laboratory tests to monitor participants' liver function was left to the treating physician's clinical judgment. The mean values and standard deviations for those tested at Week 36 are presented.
Time Frame: Week 36
Population: Participants with aspartate aminotransferase and alanine aminotransferase results at Week 36.
Measure: Mean (Standard Deviation); unit: U/liter
Arm/Group | HIV-infected Participants With Hepatitis Co-infection: AST | HIV-infected Participants With Hepatitis Co-infection: ALT
Number analyzed (Participants) | 23 | 23
U/liter | 54 (33) | 75 (87)

6. Primary Outcome: Aspartate Aminotransferase (AST) / Alanine Aminotransferase (ALT) Parameters
Description: The decision to perform aspartate aminotransferase (AST) and alanine aminotransferase (ALT) laboratory tests to monitor participants' liver function was left to the treating physician's clinical judgment. The mean values and standard deviations for those tested at Week 48 are presented.
Time Frame: Week 48
Population: Participants with aspartate aminotransferase and alanine aminotransferase results at Week 48.
Measure: Mean (Standard Deviation); unit: U/liter
Arm/Group | HIV-infected Participants With Hepatitis Co-infection: AST | HIV-infected Participants With Hepatitis Co-infection: ALT
Number analyzed (Participants) | 23 | 23
U/liter | 60 (41) | 79 (92)

7. Primary Outcome: Aspartate Aminotransferase (AST) / Alanine Aminotransferase (ALT) Parameters
Description: The decision to perform aspartate aminotransferase (AST) and alanine aminotransferase (ALT) laboratory tests to monitor participants' liver function was left to the treating physician's clinical judgment. The mean values and standard deviations for those tested at Week 60 are presented.
Time Frame: Week 60
Population: Participants with aspartate aminotransferase and alanine aminotransferase results at Week 60.
Measure: Mean (Standard Deviation); unit: U/liter
Arm/Group | HIV-infected Participants With Hepatitis Co-infection: AST | HIV-infected Participants With Hepatitis Co-infection: ALT
Number analyzed (Participants) | 23 | 23
U/liter | 55 (38) | 59 (50)

8. Primary Outcome: Aspartate Aminotransferase (AST) / Alanine Aminotransferase (ALT) Parameters
Description: The decision to perform aspartate aminotransferase (AST) and alanine aminotransferase (ALT) laboratory tests to monitor participants' liver function was left to the treating physician's clinical judgment. The mean values and standard deviations for those tested at Week 72 are presented.
Time Frame: Week 72
Population: Participants with aspartate aminotransferase and alanine aminotransferase results at Week 72.
Measure: Mean (Standard Deviation); unit: U/liter
Arm/Group | HIV-infected Participants With Hepatitis Co-infection: AST | HIV-infected Participants With Hepatitis Co-infection: ALT
Number analyzed (Participants) | 20 | 20
U/liter | 51 (36) | 50 (35)

9. Primary Outcome: Aspartate Aminotransferase (AST) / Alanine Aminotransferase (ALT) Parameters
Description: The decision to perform aspartate aminotransferase (AST) and alanine aminotransferase (ALT) laboratory tests to monitor participants' liver function was left to the treating physician's clinical judgment. The mean values and standard deviations for those tested at Week 84 are presented.
Time Frame: Week 84
Population: Participants with aspartate aminotransferase and alanine aminotransferase results at Week 84.
Measure: Mean (Standard Deviation); unit: U/liter
Arm/Group | HIV-infected Participants With Hepatitis Co-infection: AST | HIV-infected Participants With Hepatitis Co-infection: ALT
Number analyzed (Participants) | 17 | 18
U/liter | 55 (33) | 49 (27)

10. Primary Outcome: Aspartate Aminotransferase (AST) / Alanine Aminotransferase (ALT) Parameters
Description: The decision to perform aspartate aminotransferase (AST) and alanine aminotransferase (ALT) laboratory tests to monitor participants' liver function was left to the treating physician's clinical judgment. The mean values and standard deviations for those tested at Week 96 are presented.
Time Frame: Week 96
Population: Participants with aspartate aminotransferase and alanine aminotransferase results at Week 96.
Measure: Mean (Standard Deviation); unit: U/liter
Arm/Group | HIV-infected Participants With Hepatitis Co-infection: AST | HIV-infected Participants With Hepatitis Co-infection: ALT
Number analyzed (Participants) | 15 | 15
U/liter | 63 (44) | 63 (45)

11. Primary Outcome: Aspartate Aminotransferase (AST) / Alanine Aminotransferase (ALT) Parameters
Description: The decision to perform aspartate aminotransferase (AST) and alanine aminotransferase (ALT) laboratory tests to monitor participants' liver function was left to the treating physician's clinical judgment. The mean values and standard deviations for those tested at Week 108 are presented.
Time Frame: Week 108
Population: Participants with aspartate aminotransferase and alanine aminotransferase results at Week 108.
Measure: Mean (Standard Deviation); unit: U/liter
Arm/Group | HIV-infected Participants With Hepatitis Co-infection: AST | HIV-infected Participants With Hepatitis Co-infection: ALT
Number analyzed (Participants) | 18 | 19
U/liter | 47 (19) | 43 (20)

12. Primary Outcome: Aspartate Aminotransferase (AST) / Alanine Aminotransferase (ALT) Parameters
Description: The decision to perform aspartate aminotransferase (AST) and alanine aminotransferase (ALT) laboratory tests to monitor participants' liver function was left to the treating physician's clinical judgment. The mean values and standard deviations for those tested at Week 120 are presented.
Time Frame: Week 120
Population: Participants with aspartate aminotransferase and alanine aminotransferase results at Week 120.
Measure: Mean (Standard Deviation); unit: U/liter
Arm/Group | HIV-infected Participants With Hepatitis Co-infection: AST | HIV-infected Participants With Hepatitis Co-infection: ALT
Number analyzed (Participants) | 17 | 17
U/liter | 56 (30) | 65 (39)

13. Primary Outcome: Aspartate Aminotransferase (AST) / Alanine Aminotransferase (ALT) Parameters
Description: The decision to perform aspartate aminotransferase (AST) and alanine aminotransferase (ALT) laboratory tests to monitor participants' liver function was left to the treating physician's clinical judgment. The mean values and standard deviations for those tested at Week 132 are presented.
Time Frame: Week 132
Population: Participants with aspartate aminotransferase and alanine aminotransferase results at Week 132.
Measure: Mean (Standard Deviation); unit: U/liter
Arm/Group | HIV-infected Participants With Hepatitis Co-infection: AST | HIV-infected Participants With Hepatitis Co-infection: ALT
Number analyzed (Participants) | 15 | 15
U/liter | 49 (24) | 51 (31)

14. Primary Outcome: Aspartate Aminotransferase (AST) / Alanine Aminotransferase (ALT) Parameters
Description: The decision to perform aspartate aminotransferase (AST) and alanine aminotransferase (ALT) laboratory tests to monitor participants' liver function was left to the treating physician's clinical judgment. The mean values and standard deviations for those tested at Week 144 are presented.
Time Frame: Week 144
Population: Participants with aspartate aminotransferase and alanine aminotransferase results at Week 144.
Measure: Mean (Standard Deviation); unit: U/liter
Arm/Group | HIV-infected Participants With Hepatitis Co-infection: AST | HIV-infected Participants With Hepatitis Co-infection: ALT
Number analyzed (Participants) | 17 | 17
U/liter | 52 (28) | 53 (36)

15. Primary Outcome: Viral Load
Description: The decision to perform HIV-1 ribonucleic acid (RNA) tests to monitor participants' viral load was left to the treating physician's clinical judgment. The mean values and standard deviations for those tested at Baseline are presented.
Time Frame: Baseline
Population: Participants with HIV-1 RNA results at Baseline.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Number analyzed (Participants) | 24
log10 copies/mL | 3.9 (1.4)

16. Primary Outcome: Viral Load
Description: The decision to perform HIV-1 ribonucleic acid (RNA) tests to monitor participants' viral load was left to the treating physician's clinical judgment. The mean values and standard deviations for those tested at Week 4 are presented.
Time Frame: Week 4
Population: Participants with HIV-1 RNA results at Week 4.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Number analyzed (Participants) | 22
log10 copies/mL | 2.5 (0.8)

17. Primary Outcome: Viral Load
Description: The decision to perform HIV-1 ribonucleic acid (RNA) tests to monitor participants' viral load was left to the treating physician's clinical judgment. The mean values and standard deviations for those tested at Week 12 are presented.
Time Frame: Week 12
Population: Participants with HIV-1 RNA results at Week 12.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Number analyzed (Participants) | 22
log10 copies/mL | 2.0 (0.5)

18. Primary Outcome: Viral Load
Description: The decision to perform HIV-1 ribonucleic acid (RNA) tests to monitor participants' viral load was left to the treating physician's clinical judgment. The mean values and standard deviations for those tested at Week 24 are presented.
Time Frame: Week 24
Population: Participants with HIV-1 RNA results at Week 24.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Number analyzed (Participants) | 22
log10 copies/mL | 1.7 (0.4)

19. Primary Outcome: Viral Load
Description: The decision to perform HIV-1 ribonucleic acid (RNA) tests to monitor participants' viral load was left to the treating physician's clinical judgment. The mean values and standard deviations for those tested at Week 36 are presented.
Time Frame: Week 36
Population: Participants with HIV-1 RNA results at Week 36.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Number analyzed (Participants) | 22
log10 copies/mL | 1.6 (0.2)

20. Primary Outcome: Viral Load
Description: The decision to perform HIV-1 ribonucleic acid (RNA) tests to monitor participants' viral load was left to the treating physician's clinical judgment. The mean values and standard deviations for those tested at Week 48 are presented.
Time Frame: Week 48
Population: Participants with HIV-1 RNA results at Week 48.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Number analyzed (Participants) | 23
log10 copies/mL | 1.7 (0.3)

21. Primary Outcome: Viral Load
Description: The decision to perform HIV-1 ribonucleic acid (RNA) tests to monitor participants' viral load was left to the treating physician's clinical judgment. The mean values and standard deviations for those tested at Week 60 are presented.
Time Frame: Week 60
Population: Participants with HIV-1 RNA results at Week 60.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Number analyzed (Participants) | 24
log10 copies/mL | 1.7 (0.4)

22. Primary Outcome: Viral Load
Description: The decision to perform HIV-1 ribonucleic acid (RNA) tests to monitor participants' viral load was left to the treating physician's clinical judgment. The mean values and standard deviations for those tested at Week 72 are presented.
Time Frame: Week 72
Population: Participants with HIV-1 RNA results at Week 72.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Number analyzed (Participants) | 17
log10 copies/mL | 1.6 (0.2)

23. Primary Outcome: Viral Load
Description: The decision to perform HIV-1 ribonucleic acid (RNA) tests to monitor participants' viral load was left to the treating physician's clinical judgment. The mean values and standard deviations for those tested at Week 84 are presented.
Time Frame: Week 84
Population: Participants with HIV-1 RNA results at Week 84.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Number analyzed (Participants) | 18
log10 copies/mL | 1.5 (0.3)

24. Primary Outcome: Viral Load
Description: The decision to perform HIV-1 ribonucleic acid (RNA) tests to monitor participants' viral load was left to the treating physician's clinical judgment. The mean values and standard deviations for those tested at Week 96 are presented.
Time Frame: Week 96
Population: Participants with HIV-1 RNA results at Week 96.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Number analyzed (Participants) | 15
log10 copies/mL | 1.6 (0.3)

25. Primary Outcome: Viral Load
Description: The decision to perform HIV-1 ribonucleic acid (RNA) tests to monitor participants' viral load was left to the treating physician's clinical judgment. The mean values and standard deviations for those tested at Week 108 are presented.
Time Frame: Week 108
Population: Participants with HIV-1 RNA results at Week 108.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Number analyzed (Participants) | 19
log10 copies/mL | 1.6 (0.4)

26. Primary Outcome: Viral Load
Description: The decision to perform HIV-1 ribonucleic acid (RNA) tests to monitor participants' viral load was left to the treating physician's clinical judgment. The mean values and standard deviations for those tested at Week 120 are presented.
Time Frame: Week 120
Population: Participants with HIV-1 RNA results at Week 120.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Number analyzed (Participants) | 16
log10 copies/mL | 1.6 (0.4)

27. Primary Outcome: Viral Load
Description: The decision to perform HIV-1 ribonucleic acid (RNA) tests to monitor participants' viral load was left to the treating physician's clinical judgment. The mean values and standard deviations for those tested at Week 132 are presented.
Time Frame: Week 132
Population: Participants with HIV-1 RNA results at Week 132.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Number analyzed (Participants) | 15
log10 copies/mL | 1.6 (0.3)

28. Primary Outcome: Viral Load
Description: The decision to perform HIV-1 ribonucleic acid (RNA) tests to monitor participants' viral load was left to the treating physician's clinical judgment. The mean values and standard deviations for those tested at Week 144 are presented.
Time Frame: Week 144
Population: Participants with HIV-1 RNA results at Week 144.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Number analyzed (Participants) | 17
log10 copies/mL | 1.5 (0.2)

29. Primary Outcome: CD4 Cell Count
Description: The decision to perform laboratory tests to determine participants' CD4-positive (CD4+) T-lymphocyte counts was left to the treating physician's clinical judgment. The mean and standard deviation for those tested at Baseline are presented.
Time Frame: Baseline
Population: All participants with CD4+ cell count measurements at Baseline are included.
Measure: Mean (Standard Deviation); unit: CD4+ cells/μL
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Number analyzed (Participants) | 33
CD4+ cells/μL | 288 (192)

30. Primary Outcome: CD4 Cell Count
Description: The decision to perform laboratory tests to determine participants' CD4-positive (CD4+) T-lymphocyte counts was left to the treating physician's clinical judgment. The mean and standard deviation for those tested at Week 4 are presented.
Time Frame: Week 4
Population: All participants with CD4+ cell count measurements at Week 4 are included.
Measure: Mean (Standard Deviation); unit: CD4+ cells/μL
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Number analyzed (Participants) | 22
CD4+ cells/μL | 350 (165)

31. Primary Outcome: CD4 Cell Count
Description: The decision to perform laboratory tests to determine participants' CD4-positive (CD4+) T-lymphocyte counts was left to the treating physician's clinical judgment. The mean and standard deviation for those tested at Week 12 are presented.
Time Frame: Week 12
Population: All participants with CD4+ cell count measurements at Week 12 are included.
Measure: Mean (Standard Deviation); unit: CD4+ cells/μL
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Number analyzed (Participants) | 23
CD4+ cells/μL | 378 (204)

32. Primary Outcome: CD4 Cell Count
Description: The decision to perform laboratory tests to determine participants' CD4-positive (CD4+) T-lymphocyte counts was left to the treating physician's clinical judgment. The mean and standard deviation for those tested at Week 24 are presented.
Time Frame: Week 24
Population: All participants with CD4+ cell count measurements at Week 24 are included.
Measure: Mean (Standard Deviation); unit: CD4+ cells/μL
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Number analyzed (Participants) | 23
CD4+ cells/μL | 383 (211)

33. Primary Outcome: CD4 Cell Count
Description: The decision to perform laboratory tests to determine participants' CD4-positive (CD4+) T-lymphocyte counts was left to the treating physician's clinical judgment. The mean and standard deviation for those tested at Week 36 are presented.
Time Frame: Week 36
Population: All participants with CD4+ cell count measurements at Week 36 are included.
Measure: Mean (Standard Deviation); unit: CD4+ cells/μL
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Number analyzed (Participants) | 22
CD4+ cells/μL | 408 (187)

34. Primary Outcome: CD4 Cell Count
Description: The decision to perform laboratory tests to determine participants' CD4-positive (CD4+) T-lymphocyte counts was left to the treating physician's clinical judgment. The mean and standard deviation for those tested at Week 48 are presented.
Time Frame: Week 48
Population: All participants with CD4+ cell count measurements at Week 48 are included.
Measure: Mean (Standard Deviation); unit: CD4+ cells/μL
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Number analyzed (Participants) | 23
CD4+ cells/μL | 402 (239)

35. Primary Outcome: CD4 Cell Count
Description: The decision to perform laboratory tests to determine participants' CD4-positive (CD4+) T-lymphocyte counts was left to the treating physician's clinical judgment. The mean and standard deviation for those tested at Week 60 are presented.
Time Frame: Week 60
Population: All participants with CD4+ cell count measurements at Baseline are included.
Measure: Mean (Standard Deviation); unit: CD4+ cells/μL
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Number analyzed (Participants) | 24
CD4+ cells/μL | 424 (193)

36. Primary Outcome: CD4 Cell Count
Description: The decision to perform laboratory tests to determine participants' CD4-positive (CD4+) T-lymphocyte counts was left to the treating physician's clinical judgment. The mean and standard deviation for those tested at Week 72 are presented.
Time Frame: Week 72
Population: All participants with CD4+ cell count measurements at Week 72 are included.
Measure: Mean (Standard Deviation); unit: CD4+ cells/μL
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Number analyzed (Participants) | 18
CD4+ cells/μL | 431 (235)

37. Primary Outcome: CD4 Cell Count
Description: The decision to perform laboratory tests to determine participants' CD4-positive (CD4+) T-lymphocyte counts was left to the treating physician's clinical judgment. The mean and standard deviation for those tested at Week 84 are presented.
Time Frame: Week 84
Population: All participants with CD4+ cell count measurements at Week 84 are included.
Measure: Mean (Standard Deviation); unit: CD4+ cells/μL
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Number analyzed (Participants) | 18
CD4+ cells/μL | 405 (170)

38. Primary Outcome: CD4 Cell Count
Description: The decision to perform laboratory tests to determine participants' CD4-positive (CD4+) T-lymphocyte counts was left to the treating physician's clinical judgment. The mean and standard deviation for those tested at Week 96 are presented.
Time Frame: Week 96
Population: All participants with CD4+ cell count measurements at Week 96 are included.
Measure: Mean (Standard Deviation); unit: CD4+ cells/μL
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Number analyzed (Participants) | 14
CD4+ cells/μL | 503 (237)

39. Primary Outcome: CD4 Cell Count
Description: The decision to perform laboratory tests to determine participants' CD4-positive (CD4+) T-lymphocyte counts was left to the treating physician's clinical judgment. The mean and standard deviation for those tested at Week 108 are presented.
Time Frame: Week 108
Population: All participants with CD4+ cell count measurements at Week 108 are included.
Measure: Mean (Standard Deviation); unit: CD4+ cells/μL
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Number analyzed (Participants) | 18
CD4+ cells/μL | 581 (303)

40. Primary Outcome: CD4 Cell Count
Description: The decision to perform laboratory tests to determine participants' CD4-positive (CD4+) T-lymphocyte counts was left to the treating physician's clinical judgment. The mean and standard deviation for those tested at Week 120 are presented.
Time Frame: Week 120
Population: All participants with CD4+ cell count measurements at Week 120 are included.
Measure: Mean (Standard Deviation); unit: CD4+ cells/μL
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Number analyzed (Participants) | 15
CD4+ cells/μL | 565 (256)

41. Primary Outcome: CD4 Cell Count
Description: The decision to perform laboratory tests to determine participants' CD4-positive (CD4+) T-lymphocyte counts was left to the treating physician's clinical judgment. The mean and standard deviation for those tested at Week 132 are presented.
Time Frame: Week 132
Population: All participants with CD4+ cell count measurements at Week 132 are included.
Measure: Mean (Standard Deviation); unit: CD4+ cells/μL
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Number analyzed (Participants) | 15
CD4+ cells/μL | 502 (259)

42. Primary Outcome: CD4 Cell Count
Description: The decision to perform laboratory tests to determine participants' CD4-positive (CD4+) T-lymphocyte counts was left to the treating physician's clinical judgment. The mean and standard deviation for those tested at Week 144 are presented.
Time Frame: Week 144
Population: All participants with CD4+ cell count measurements at Week 144 are included.
Measure: Mean (Standard Deviation); unit: CD4+ cells/μL
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Number analyzed (Participants) | 17
CD4+ cells/μL | 525 (226)

ADVERSE EVENTS:
Time Frame: Investigators were instructed to report adverse events throughout the study (up to 3 years).
Arm/Group | HIV-infected Participants With Hepatitis Co-infection
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 1/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIV-infected Participants With Hepatitis Co-infection (N=33)
antiviral drug level above therapeutic (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.